CLINICAL TRIAL: NCT01261520
Title: Promoting Adherence to Mammography Use in Chinese Women
Brief Title: Chinese Women and Mammography Screening
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Judy Wang, Assistant Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GU 2005-167; MRSGT-05-104-01-CPPB (Other Grant/Funding Number: American Cancer Society); R03CA117552 (NIH)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Study Chinese Women Who Have Not Adhered to American Cancer Society Mammography Screening Guideline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Culturally-tailored video (Other): The culturally-tailored video was designed to focus on Chinese women's cultural health beliefs and align with Chinese customs, norms, and values, which includes two segments: 1) a soap-opera and 2) recommendation from a Chinese female physician.
  Interventions: Behavioral: Culturally-tailored video

INTERVENTIONS:
Behavioral: Culturally-tailored video — A 18 minute DVD made in Chinese language (i.e. Mandarin and Cantonese)

SUMMARY:
This study examined whether a culturally-tailored video has a greater impact on increasing mammography use in Chinese American women and improving barriers to mammography screening compared to a generic, non-tailored video and a printed fact sheet (control group).

DETAILED DESCRIPTION:
This study examined the efficacy of a culturally-tailored video in increasing mammography use among non-adherent Chinese women (vs. a generic video and control fact sheet). A total of 671 Chinese American women from metropolitan Washington, DC and New York city were enrolled to participate in this study. The majority of participants were recruited from on-site community events and some were recruited through public advertisement and referrals. Participants who completed baseline assessment were randomized to one of the three groups: 1) viewing an 18-minute cultural video, 2) viewing an 18-minute generic video, and 3) reading a fact sheet (control group). Participants were interviewed twice after intervention:1) process evaluation 2-4 weeks post intervention regarding participants' feedback on the materials and repeated key measures of knowledge, cultural views, and health beliefs and 2) outcome evaluation six-months post intervention that assesses actual receipt of mammography use.

ELIGIBILITY:
Inclusion Criteria:

* Chinese American women had not had a mammography in the past 12 months
* Chinese American women had no personal history of breast cancer
* Chinese American women had no mammogram scheduled when enrolled

Exclusion Criteria:

* Non-Chinese Women
* Regular mammography users

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2005-07; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Receipt of mammography screening | six month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Judy H Wang, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Cancer Control Program, Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Wang JH, Mandelblatt JS, Liang W, Yi B, Ma IJ, Schwartz MD. Knowledge, cultural, and attitudinal barriers to mammography screening among nonadherent immigrant Chinese women: ever versus never screened status. Cancer. 2009 Oct 15;115(20):4828-38. doi: 10.1002/cncr.24517. PMID 19645031
- [Derived] Wang JH, Sheppard VB, Liang W, Ma GX, Maxwell AE. Recruiting Chinese Americans into cancer screening intervention trials: strategies and outcomes. Clin Trials. 2014 Apr;11(2):167-77. doi: 10.1177/1740774513518849. Epub 2014 Feb 24. PMID 24567288